CLINICAL TRIAL: NCT00771576
Title: PET Scan Imaging of Pancreatic Beta Cell Mass With DTBZ
Brief Title: PET Scan Imaging of Beta Cell Mass
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAB0002
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetes; Obesity
Keywords: Diabetes Mellitus; T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A. Healthy Controls: subjects w/ predicted normal BCM (healthy, normalweight, nondiabetic individuals who have stimulated insulin and cpeptide levels within the normal range);
- B. Longstanding T1D: subjects with predicted reduced beta cell mass (subjects with established T1DM who have low or not measurable stimulated insulin and c peptide levels);
- C. Obese Subjects: subjects with predicted increased beta cell mass (euglycemic obese subjects with fasting hyperinsulinemia).

SUMMARY:
The investigators hypothesize that PET scans will be able to differentiate between normal, reduced or increased BCM in human subjects. Subjects with normal BCM will be recruited from among normal weight nondiabetic people with plasma insulin levels within the normal range. Subjects with predicted reduced BCM will be recruited from among patients with T1DM who have with low or not measurable insulin levels. If results from the nondiabetic subjects and the subjects with T1DM are found to differ significantly, subjects with increased BCM will be recruited from among patients with hyperinsulinemia including those with obesity and the metabolic syndrome. PET scan measurements of the pancreas will be obtained and compared in people predicted, on the basis of biochemical testing, to have normal or reduced, or increased BCM.

DETAILED DESCRIPTION:
An important determinant of progression to diabetes is beta cell mass (BCM). Measurement of plasma insulin has been used as a surrogate marker but insulin levels often do not correlate well with beta cell mass and development of means to assess BCM would provide an important endpoint. For example, high-risk individuals could be monitored prior to onset of diabetes or patients could be monitored prospectively to determine the progression of their disease and response to therapy.

Both Type 1 diabetes mellitus (T1DM) and Type 2 diabetes mellitus (T2DM) develop when there is impaired insulin production. The amount of insulin that can be produced, the amount of insulin producing beta cells in the pancreas and level of insulin and glucose in the blood are, however, imperfectly correlated. The development of a reliable method to noninvasively quantitate the beta cell mass (BCM) would be of great benefit by providing an important endpoint for the development of new treatments of T1DM and T2DM. The investigators have previously identified a specific marker on islet cells called vesicular monoamine transporter 2 (VMAT2) that they now propose to use in positron emission tomography (PET) scanning to determine islet cell mass. This radioligand, [11C] Dihydrotetrabenazine (DTBZ), has been used previously in human subjects in clinical trials evaluating PET scanning of the brain in patients with bipolar illness and schizophrenia compared to healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must meet all of the following inclusion criteria:

1. Informed consent obtained from participants
2. Age 18-45 years
3. Healthy non-diabetic subjects will have normal fasting blood sugar (<100 mg/dl), body mass index (BMI) 18.5-24.9, no history of type 2 diabetes in first degree relative
4. Type 1 diabetes defined by: American Diabetes Association (ADA) criteria or judgment of physician; diabetes onset younger than age 18, duration >5 - years, BMI 18.5-24.9. Insulin dose <0.8 units/kg/day. Fasting c-peptide < 0.1 ng/ml
5. Obese hyper-insulinemic subjects will have BMI > 30 and fasting insulin>20 and c-peptide> 4.6 ng/ml and normal fasting blood sugar <100 mg/dl.
6. Able to tolerate PET imaging: not claustrophobic, able to lie supine for 1.5 hours
7. Normal liver and renal function tests including normal spot urine microalbumin /creatinine; normal CBC including hematocrit >31.8% in women, >36.7% in men, white blood cell (WBC) count >3.4 K/mm3 and platelet count >162 K/mm3
8. Adequate collateral circulation in the wrist as assessed by Allen Test.

Exclusion Criteria:

Potential participants must not have any of the following exclusion criteria:

1. Previous or current treatment with drugs influencing beta cell function or insulin sensitivity (e.g. oral hypoglycemic agents, glucocorticoids); or with antipsychotic, antianxiety, or antidepressant medications (eg monoamine oxidase (MAO) inhibitors, 5-hydroxytryptamine (5-HT) inhibitors, tricyclic antidepressants); or treatment with reserpine; or treatment with beta2receptor agonists (eg, terbutaline); or treatment with anticoagulant medication.
2. History of movement disorder such as Parkinson's Disease or Huntington's Disease
3. History of or psychiatric illness such as depression, bipolar disease, anxiety or schizophrenia.
4. If a female of childbearing age, currently pregnant, breastfeeding or not using a form of birth control
5. Previous or current use of cocaine, methamphetamine, ecstasy
6. Current daily intake of caffeine >500 mg/day (>45 cups of coffee; >10 12oz cans of soda)
7. Current history of cigarette smoking
8. Consumption of more than 1 alcoholic drink per day
9. Evidence of chronic infection
10. History of malignancy
11. Any prior participation in other research protocols within the past year that involve radiation, with the exception of plain radiography studies (i.e., chest xrays).
12. Medical implant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Potential subjects with diabetes will be recruited from among the patients cared for at the Naomi Berrie Diabetes Center. Nondiabetic subjects will either be referred by their physicians or by word of mouth. Primary care physicians will be made aware of the study by fliers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2012-06-13 (Actual)

PRIMARY OUTCOMES:
Pancreas [11C] DTBZ binding | Once

CONTACTS AND LOCATIONS:
Overall Officials: PAUL E HARRIS, Ph.D., Study Director — Columbia University; Robin S Goland, M.D., Principal Investigator — Columbia University; Ronald Van Heertum, M.D., Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Naomi Berrie Diabetes Cener, New York, New York
  - Kreitchman PET Center Columbia University Medical Center, New York, New York

REFERENCES:
- [Background] Souza F, Simpson N, Raffo A, Saxena C, Maffei A, Hardy M, Kilbourn M, Goland R, Leibel R, Mann JJ, Van Heertum R, Harris PE. Longitudinal noninvasive PET-based beta cell mass estimates in a spontaneous diabetes rat model. J Clin Invest. 2006 Jun;116(6):1506-13. doi: 10.1172/JCI27645. Epub 2006 May 18. PMID 16710474
- [Background] Simpson NR, Souza F, Witkowski P, Maffei A, Raffo A, Herron A, Kilbourn M, Jurewicz A, Herold K, Liu E, Hardy MA, Van Heertum R, Harris PE. Visualizing pancreatic beta-cell mass with [11C]DTBZ. Nucl Med Biol. 2006 Oct;33(7):855-64. doi: 10.1016/j.nucmedbio.2006.07.002. PMID 17045165
- [Background] Murthy R, Harris P, Simpson N, Van Heertum R, Leibel R, Mann JJ, Parsey R. Whole body [11C]-dihydrotetrabenazine imaging of baboons: biodistribution and human radiation dosimetry estimates. Eur J Nucl Med Mol Imaging. 2008 Apr;35(4):790-7. doi: 10.1007/s00259-007-0648-2. Epub 2007 Dec 4. PMID 18060547